CLINICAL TRIAL: NCT07005713
Title: A Phase 1b, Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of Multiple- Ascending Doses of BGB-16673 in Patients With Chronic Spontaneous Urticaria
Brief Title: A Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of Multiple-Ascending Doses of BGB-16673 in Adults With Chronic Spontaneous Urticaria
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: BeiGene (Industry)
Responsible Party: Sponsor
Organization: BeOne Medicines (Industry)
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: BGB-16673-107
Record Dates: First submitted 2025-05-22; First posted 2025-06-05 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Chronic Spontaneous Urticaria
MeSH Terms: conditions — Chronic Urticaria

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BGB-16673 (Experimental): Participants will receive BGB-16673 orally
  Interventions: Drug: BGB-16673
- Placebo (Placebo Comparator): Participants will receive placebo orally for 28 days and then crossover to receive BGB-16673.
  Interventions: Drug: BGB-16673; Drug: Placebo

INTERVENTIONS:
Drug: BGB-16673 — Administered orally
Drug: Placebo — Administered orally
  Arms: Placebo

SUMMARY:
This study is a Phase 1b, randomized, double-blind, placebo-controlled study to evaluate the safety, tolerability, pharmacokinetics (PK), and pharmacodynamics of multiple-ascending doses of BGB-16673 in adults with chronic spontaneous urticaria (CSU).

ELIGIBILITY:
Inclusion Criteria:

* Participants must be diagnosed with chronic spontaneous urticaria (CSU) for ≥ 6 months before randomization.
* The presence of itch and hives for ≥6 consecutive weeks at any time prior to randomization despite the use of second-generation H1-antihistamines
* UAS7≥16 and HSS7≥8 during the 7 days before randomization
* Participants must not have had any missing UAS7 entry (ISS7 and HSS7) during the 7 days before randomization
* Presence of hives must have been documented within 3 months before randomization

Exclusion Criteria:

* Participants who have a clearly defined, predominating or sole trigger for their chronic urticaria (chronic inducible urticaria), including urticaria factitia (symptomatic dermographism) or cold, heat, solar, pressure, delayed pressure, aquagenic, cholinergic, or contact urticaria.
* Other diseases with symptoms of urticaria or angioedema
* Any other skin disease associated with chronic itching that might influence in the investigators opinion the study evaluations and results, eg, atopic dermatitis, bullous pemphigoid, dermatitis herpetiformis, senile pruritus, or psoriasis.
* Any uncontrolled disease state, including asthma or inflammatory bowel disease where flares are commonly treated with oral or parenteral corticosteroids.
* Significant bleeding risk or coagulopathy.
* Prior exposure to any BTK inhibitors or protein degraders.

NOTE: Other protocol defined Inclusion/Exclusion criteria may apply.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2025-07-19 (Actual); Primary Completion 2026-04-17 (Estimated); Study Completion 2026-04-17 (Estimated)

PRIMARY OUTCOMES:
Number of participants with adverse events (AEs) | Up to approximately 4 months
  Number of participants with treatment-emergent adverse events (TEAEs) and serious adverse events (SAEs), including findings from laboratory tests and electrocardiogram results.
Maximum observed plasma concentration (Cmax) of BGB-16673 | Up to approximately 10 weeks
Minimum observed plasma concentration (Cmin) of BGB-16673 | Up to approximately 10 weeks
Time to reach maximum observed plasma concentration (Tmax) of BGB-16673 | Up to approximately 10 weeks
Apparent terminal elimination half life (t1/2) of BGB-16673 | Up to approximately 10 weeks
Area under the curve (AUC) of BGB-16673 | Up to approximately 10 weeks
Apparent oral clearance (CL/F) of BGB-16673 | Up to approximately 10 weeks
Apparent volume of distribution (Vz/F) of BGB-16673 | Up to approximately 10 weeks
Accumulation Ratio of AUC for BGB-16673 | Up to approximately 10 weeks
Accumulation Ratio of Cmax for BGB-16673 | Up to approximately 10 weeks

SECONDARY OUTCOMES:
Change from Baseline in Weekly Urticaria Activity Score (UAS7) | Baseline and up to approximately 3 months
  The UAS7 consists of an assessment of both hives and itch severity to provide a measure of disease activity. The UAS7 is the sum of the weekly Hives Severity Score (HSS7) and the weekly Itch Severity Score (ISS7) and ranges between 0 and 42. A UAS7 score of 0 signifies that the patient is symptom free, and high UAS7 scores indicate severe symptoms.
Change from baseline in weekly Itch Severity Score (ISS7) | Baseline and up to approximately 3 months
  The Itch Severity Score (ISS) is a measure of itching. Daily scores range from 0 (no itching) to 3 (intense itching). The ISS7 is a weekly score derived by adding up the daily ISS scores of the past 7 days and ranges from 0 to 21.
Change from baseline in weekly Hives Severity Score (HSS7) | Baseline and up to approximately 3 months
  The Hives Severity Score (HSS) is a measure of the number of hives present recorded by the participant. Daily scores range from 0 (no hives) to 3 (intense/severe hives). HSS7 is the sum of the daily HSS scores over the past 7 days and ranges from 0 to 21.
Change from baseline in weekly Angioedema Activity Score (AAS7) | Baseline and up to approximately 3 months
  The Angioedema Activity Score (AAS) is a validated tool designed and verified to measure disease activity, assess response to treatment, and optimize the treatment plan for patients with recurrent angioedema. Responses are filled out prospectively and daily, evaluating five main factors related to angioedema: duration, physical discomfort caused, impact on daily activities, effect on appearance, and overall severity, each scored between 0 and 3. Daily AAS scores can range daily from 0 to 15, and weekly (AAS7) from 0 to 105. Higher AAS scores indicate frequent and severe attacks. Lower scores indicate well-controlled symptoms.
Change from baseline in 7-day recall period version of the Urticaria Control Test (UCT7) | Baseline and up to approximately 3 months
  UCT7 is a validated questionnaire used to measure the quality of life of patients with chronic urticaria and angioedema. It contains 4 questions, each of which inquires about the extent of impairment in the previous 7 days, with 5 options for answers ranging from "not at all" to "very much." The first question asks about the frequency of all symptoms combined (itching, hives, and/or swelling). The second question asks about the overall impact on quality of life. The third question asks how often treatment has been insufficient to control symptoms, and the final question asks about how well the disease has been controlled. Answers are scored from 0 to 4 (the total score will range from 0 to 16), with higher scores representing milder and better-controlled urticaria and angioedema. The recall period for this questionnaire is 7 days.
Percentage of participants with complete absence of hives and itch, assessed as UAS7 = 0 | Up to approximately 3 months
Percentage of participants with UAS7 ≤ 6 response | Up to approximately 3 months
Levels of Bruton tyrosine kinase (BTK) protein | Up to approximately 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — BeiGene
Locations (8):
- China (8):
  - Peking University Third Hospital, Beijing, Beijing Municipality
  - The First Affiliated Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality
  - Dermatology Hospital of Southern Medical University, Guangzhou, Guangdong
  - Union Hospital of Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei
  - Xiangya Hospital of Central South University, Changsha, Hunan
  - Chengdu Second Peoples Hospital, Chengdu, Sichuan
  - Hangzhou First Peoples Hospital, Hangzhou, Zhejiang
  - The First Affiliated Hospital of Wenzhou Medical University, Wenzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: Yes
BeiGene shares data on completed studies responsibly and provides qualified scientific and medical researchers access to data and supporting documentation for clinical trials in dossiers for medicines and indications after submission and approval in the United States, China, and Europe. Clinical trials supporting subsequent local approvals, new indications, or combination products are eligible for sharing once corresponding regulatory approvals are achieved.
  BeiGene shares data only when permitted by applicable data privacy and security laws and regulations, when it is feasible to do so without compromising the privacy of study participants, and other considerations.
  Qualified researchers with appropriate competencies who are engaged in novel scientific research may submit a request for participant-level data with a research proposal for BeiGene review. Research teams must include a biostatistician and sign a Data Sharing Agreement prior to receiving access to clinical trial data.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: See plan description
Access Criteria: See plan description
URL: https://beigene.com/science/clinical-trials/